CLINICAL TRIAL: NCT00819312
Title: A Multicenter, Open-label, Single-arm Study to Investigate the Efficacy and Safety of the Oral Contraceptive YAZ (20 μg Ethinylestradiol, 3 mg Drospirenone) for 13 Cycles in 670 Healthy Chinese Female Volunteers.
Brief Title: YAZ, Oral Contraceptive Registration in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 91619; 311041 (Other: company internal)
Record Dates: First submitted 2009-01-05; First posted 2009-01-08 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Contraception
Keywords: Contraceptives,; Oral Hormonal;; Contraceptive Methods;; Female
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Active Comparator)
  Interventions: Drug: YAZ (SH T00186, BAY86-5300)

INTERVENTIONS:
Drug: YAZ (SH T00186, BAY86-5300) — 20ug ethinylestradiol, 3mg drospirenone, tablet, orally, opd

SUMMARY:
The purpose of this study is to evaluate the effectiveness in terms of prevention of pregnancy and safety of the oral contraceptive YAZ in healthy Chinese women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between 18 and 45 requesting oral contraception.
* Smokers may not exceed 30 years of age.

Exclusion Criteria:

* The use of steroidal oral contraceptives , or any drug that could alter oral contraception metabolism will be prohibited during the study.
* Pregnancy, lactation (less than 3 menstrual cycles since delivery, abortion or lactation before start of treatment)
* Menstrual disorders suspicious of ovarian failure (e.g. oligomenorrhea, amenorrhea, hypomenorrhea
* Any disease or condition that may worsen under hormonal treatment
* Other contraceptive methods such as sterilization or IUD/IUS
* Substantial overweight (BMI > 30 kg/m2).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 675 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the number of unintended pregnancies as measured by the Pearl Index (PI) during 13 cycles of treatment. | 13 cycles (1 cycle= 28 days)

SECONDARY OUTCOMES:
Bleeding pattern indices | 13 cycles
Cycle control parameters | 13 cycles
Adverse events | Whole study period
Laboratory tests | Whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- China (11):
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Nanjing, Jiangsu
  - Yangzhou, Jiangsu
  - Shenyang, Liaoning
  - Jinan, Shandong
  - Xi’an, Shanxi
  - Chengdu, Sichuan
  - Beijing
  - Chongqing
  - Shanghai
- Hong Kong, Hong Kong